CLINICAL TRIAL: NCT03546218
Title: Immediate Effect of Positive-word Stimuli on the Limits of Stability During Multi-direction Reach Operation in Standing Position: A Randomized Controlled Superiority Trial
Brief Title: Effect of Positive-word Stimuli on the Limits of Stability During Multi-direction Reach Operation in Standing Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kibi International University (Other)
Responsible Party: Principal Investigator, Kazuki Hirao, PhD, OT, Assistant Professor, Kibi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-16
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (SPSRS) (Experimental): Participants watch motion picture using an application that displays positive-word stimuli.
  Interventions: Device: Smartphone Application (SPSRS)
- Smartphone Application (YouTube) (Active Comparator): Participants will watch the same motion picture as the experimental group. However, a positive-word stimulus does not appear in the motion picture.
  Interventions: Device: Smartphone Application (YouTube)

INTERVENTIONS:
Device: Smartphone Application (SPSRS) — Participants use application on iPhone and watch videos showing positive-word stimuli. This application repeats positive-word stimuli every 5 seconds.
  The participants watch 3-minute motion picture displaying positive-word stimuli.
  Arms: Smartphone Application (SPSRS)
Device: Smartphone Application (YouTube) — Participants will watch the same motion picture as the experimental group. However, a positive-word stimulus does not appear in the motion picture.
  Arms: Smartphone Application (YouTube)

SUMMARY:
The purpose of the study was to examine the immediate effect of positive-word stimuli on the limits of stability during multi-direction reach operation in standing position in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 24 years of age
* Males and Females

Exclusion Criteria:

* Person with physical disability that is enough to interfere with daily life

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Multi-Directional Reach Test | Baseline and immediately after the intervention protocol
  The limits of stability during multi-direction reach operation in standing position

CONTACTS AND LOCATIONS:
Locations (1):
- Kibi International University, Takahashi, Okayama-ken, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azukizawa K, Hirose K, Morigami Y, Higashi N, Uchida H, Hirao K. Positive-word stimuli via a smartphone application have no immediate-term effects on multi-directional reach ability in standing position: a randomized controlled trial. Ann Med. 2021 Dec;53(1):1402-1409. doi: 10.1080/07853890.2021.1968483. PMID 34414832